CLINICAL TRIAL: NCT01255280
Title: Behavioral Activation and HIV Risk Reduction for MSM With Crystal Methamphetamine Abuse
Brief Title: Behavioral Activation and HIV Risk Reduction for Men Who Have Sex With Men With Crystal Meth Abuse
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Fenway Community Health (Other)
Responsible Party: Principal Investigator, Matthew James Mimiaga, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3293841
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Crystal Methamphetamine Abuse; Crystal Methamphetamine Dependence
Keywords: Crystal methamphetamine abuse; Crystal methamphetamine dependence; Sexual risk behavior; Men who have sex with men (MSM); Behavioral activation
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Information, Motivation, Behavioral skills (Active Comparator): The comparison condition will only receive the two IMB risk reduction sessions. The intervention will begin with modules that focus directly with sexual risk reduction practices. It will begin with a discussion of one's sexual history, sexual risk limits, and barriers (e.g., motivation or skills) to staying in their sexual risk limits. This session will also involve a Q&A discussion and the use of a fact sheet regarding HIV acquisition risk behaviors (information). The next session will involve motivational interviewing and the formulation of an individualized behavioral skills plan as needed.
  Interventions: Behavioral: Information, Motivation, Behavioral skills change approach to sexual risk reduction
- Behavioral Activation Therapy and Risk Reduction Counseling (Experimental): This intervention is given to patients in the experimental condition only and is comprised of 10 sessions-1 baseline session focused on orienting and rationale, 2 focused on risk reduction (consistent with the IMB model: information, motivation, and behavioral skills), 6 incorporating behavioral activation therapy/risk reduction counseling, and 1 final session on relapse prevention. Each session will last approximately fifty minutes in length; and will also involve a review of the previous materials,and hence the behavioral activation approach will be woven back into the risk reduction content.
  Interventions: Behavioral: Behavioral Activation Therapy and Risk Reduction Counseling (BAT-RR)

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy and Risk Reduction Counseling (BAT-RR) — This intervention is given to patients in the experimental condition only and is comprised of 10 sessions.
  Arms: Behavioral Activation Therapy and Risk Reduction Counseling
Behavioral: Information, Motivation, Behavioral skills change approach to sexual risk reduction — The comparison condition will only receive the two IMB risk reduction sessions.
  Arms: Information, Motivation, Behavioral skills

SUMMARY:
The purpose of this study is to research a new behavioral treatment to reduce sexual risk-taking in men who have sex with men (MSM) who abuse crystal methamphetamine (crystal meth), and are at risk for HIV acquisition. This study proposes using a treatment based on our original pilot study that incorporates risk reduction and behavioral activation therapy. In order to help learn what types of treatment programs best help individuals who abuse crystal meth and engage in sexual risk-taking, we will compare our treatment to a control group. The treatment group will receive therapy incorporating behavioral risk reduction counseling with behavioral activation therapy to treat depression, helping individuals reengage in their life. The control group will receive the risk reduction counseling without the behavioral activation therapy. The current study hopes to explore the efficacy of this previous developed treatment in a two-arm pilot randomized controlled trial.

DETAILED DESCRIPTION:
1. To estimate, in a two-arm pilot randomized controlled trial (RCT), the effect size of the proposed intervention on reductions in sexual risk taking and crystal meth use. The primary outcome is the number of unprotected anal sex acts and a secondary outcome is reduction in crystal meth use episodes over the follow up period.
2. To explore the degree to which improvements in sexual risk taking are associated with the conceptual mediators of the effects of the intervention: reductions in crystal meth use and increases in pleasurable (but safe) activities, BAT skills, use of risk reduction skills, and reductions in depressed mood.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Self-reports as a man who has sex with men
* HIV-uninfected and verifies serostatus at baseline (HIV antibody testing and positive tests will be confirmed by Western Blots; see Human Subjects for operational aspects)
* Meets DSM-IV diagnostic criteria for crystal meth abuse/dependence
* Self reported unprotected anal intercourse-receptive or insertive-with a non-monogamous male sexual partner, while concurrently using crystal meth (use of meth must be a few hours prior to, or during, sex) in the prior three months

Exclusion Criteria:

* Unable to provide informed consent due to severe mental or physical illness, or substance intoxication at the time of interview
* Has lived in the greater Boston area for three months or less (as a means to enhance participant retention)
* Discovery of active suicidal ideation at the time of interview (these patients will be referred immediately for treatment, but may join the study when this is resolved)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in sexual risk | Baseline and three months post-treatment; baseline and six months post-treatment
  We will ask about number of unprotected and protected insertive and receptive anal, vaginal and oral sex acts with male and female sex partners separately for HIV seropositive, seronegative, and partners of unknown HIV status with questions from measures used in previous studies. We will use this to calculate the ratio of protected to unprotected acts, by serostatus partner, and by whether or not crystal meth was being used before or during sex. Baseline and three and six-month follow-up assessments will assess sexual risk taking in the previous 3-months to the assessment being completed.

SECONDARY OUTCOMES:
Change in crystal methamphetamine use | Baseline and three months post-treatment; baseline and six months post-treatment
  For the present study, we will administer relevant sections of the Drug and Alcohol sections of the NIDA-CTN Addictions Severity Index Lite (ASI-Lite). We will use this methodology to determine the number of days of drug use, specifically crystal meth, and the number of distinct crystal meth episodes between study assessment visits (i.e., separate crystal meth binges).In addition to the ASI-Lite, we will also collect participant self-report measures of substance use via the ACASI. We have adapted and will also use the CDC's National HIV Behavioral Surveillance Survey, MSM cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mimiaga, ScD, Principal Investigator — Fenway Community Health and Massachusetts General Hospital/Harvard Medical School
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rajasingham R, Mimiaga MJ, White JM, Pinkston MM, Baden RP, Mitty JA. A systematic review of behavioral and treatment outcome studies among HIV-infected men who have sex with men who abuse crystal methamphetamine. AIDS Patient Care STDS. 2012 Jan;26(1):36-52. doi: 10.1089/apc.2011.0153. Epub 2011 Nov 9. PMID 22070609